CLINICAL TRIAL: NCT04903210
Title: Pilot Study of Nicotinamide Mononucleotide Supplementation in Patients With Hypertension
Brief Title: Nicotinamide Mononucleotide in Hypertensive Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Jun Tao, Prof., First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NMNHTN-001
Record Dates: First submitted 2021-05-21; First posted 2021-05-26 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2021-05

CONDITIONS: Hypertension
Keywords: Hypertension; β-nicotinamide mononucleotide; Vascular function; Blood pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Study biostatistician will be blinded to group (NMN vs. controls)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NMN group (Experimental): NMN10000 WRIGHT LIFE® + lifestyle modification.
  Interventions: Dietary Supplement: Nicotinamide mononucleotide supplied as 400mg capsule; Behavioral: Lifestyle modification
- Control group (Other): Lifestyle modification only.
  Interventions: Behavioral: Lifestyle modification

INTERVENTIONS:
Dietary Supplement: Nicotinamide mononucleotide supplied as 400mg capsule — NMN10000 WRIGHT LIFE® + lifestyle modification NMN10000 WRIGHT LIFE®: 800mg, qd, for two months. Lifestyle modification: intake 1400-1600 kcal/day: 54% carbohydrates, 24% proteins, 22% lipids, 108 mg cholesterol, 35 g fiber; avoid smoking and alcohol consumption; performing aerobic activity 4 days per week such as 45 min on a stationary bicycle.
  Arms: NMN group
Behavioral: Lifestyle modification — Lifestyle modification: intake 1400-1600 kcal/day: 54% carbohydrates, 24% proteins, 22% lipids, 108 mg cholesterol, 35 g fiber; avoid smoking and alcohol consumption; performing aerobic activity 4 days per week such as 45 min on a stationary bicycle.

SUMMARY:
Cardiovascular and cerebrovascular diseases are most terrible killers endangering the health of Chinese residents, and hypertension is the most important risk factor. Hypertension related vascular function and structural damage are the common pathological basis and initiation of cardiovascular and cerebrovascular disease. Therefore, reducing blood pressure and delaying or reversing vascular injury is an effective way to treat hypertension and prevent cardiovascular disease. NAD+ (nicotinamide adenine dinucleotide) is a coenzyme of many kinds of dehydrogenases in the body, and is an essential molecule in the basic process of life support. The latest research found that with the growth of age, the level of NAD+ is decreasing, and increasing the content of NAD+ can prolong the life of multiple species including human. NMN (β - nicotinamide mononucleotide) is a natural NAD+ precursor in cells. Recent clinical trials found that NMN supplementation can effectively improve the level of NAD+ in cells, delay aging, improve the metabolic process of cells without adverse reactions. However, the effect of NMN supplementation on reducing blood pressure and protecting vascular endothelial function has not been reported. Therefore, this study aims to focus on hypertension, a major chronic disease, and to observe the effects of NMN supplementation on vascular function and blood pressure in patients with hypertension, so as to provide a new treatment strategy for hypertension and associated vascular injury.

ELIGIBILITY:
Inclusion Criteria:

* Mild essential hypertensive patients (BP ranged from 130/80 to 159/99 mmHg).
* Ability to undergo Study procedures.
* Willingness/ability to provide informed consent.

Exclusion Criteria:

* Participants with secondary hypertension.
* Participants suffering from diabetes mellitus, coronary heart disease, peripheral vascular disease, acute or chronic liver disease, renal insufficiency, malignancies, infectious disease, or using non-steroidal anti-inflammatory drugs, steriods, vasoactive agents.
* Known allergies to niacin or nicotinamide.
* Receiving certain concurrent supplements.
* Women who are currently pregnant or who wish to become pregnant over the course of the study follow-up or who are at suckling period.
* Unwillingness/inability to provide informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-06-20 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Effect of NMN on flow mediated dilation (FMD) | Up to 2 month
  Change of FMD between NMN-treated participants and non-NMN-treated participants
Effect of NMN on brachial-ankle pulse wave velocity (baPWV) | Up to 2 month
  Change of baPWV between NMN-treated participants and non-NMN-treated participants

SECONDARY OUTCOMES:
Effect of NMN on blood pressure | Up to 2 month
  Change of systolic blood pressure and diastolic blood pressure between NMN-treated participants and non-NMN-treated participants
Effect of NMN on PBMC NAD+ levels | Up to 2 month
  Change of peripheral blood mononuclear cells NAD+ levels between NMN-treated participants and non-NMN-treated participants
Effect of NMN on sleep quality | Up to 2 month
  Change of the scores of Pittsburgh Sleep Quality Index (PSQI). The final score ranges from 0 to 21. The higher the score, the worse the sleep quality.
Incidence of Treatment Adverse Events | Up to 2 month
  Adverse Events

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital,Sun Yat-sen University, Guangzhou, Guangdong, China